CLINICAL TRIAL: NCT01016938
Title: Dynamic MRI for Lung Tumor Motion and Lung Function
Brief Title: Dynamic Magnetic Resonance Imaging (MRI) for Lung Tumor Motion and Lung Function (GCC 0943)
Status: Completed | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Department of Radiation Oncology, Principal Investigator, University of Maryland, Baltimore
Other Study IDs: HP-00043875
Record Dates: First submitted 2009-11-19; First posted 2009-11-20 (Estimated); Results first posted 2016-05-18 (Estimated); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Group I: This is a pilot study and there is only one group.

SUMMARY:
Radiation treatment for each patient with cancer is designed based on CT scans. We know that tumors in the chest and abdomen move when you breathe. Because of this, there can be differences between planned treatment and the treatment actually delivered to the body. Usually with radiation a safety margin is added to ensure that radiation hits the entire tumor. This can damage healthy parts of the body because the exact location of the tumor is unknown.

Magnetic resonance imaging (MRI) is a painless and safe diagnostic procedure that uses a powerful magnet and radio waves to produce detailed images of the body's organs and structures, without the use of X-rays or other radiation.

The research doctors are studying to see if the position of a tumor can be tracked using MRI scans and tracking sensors placed on the skin. MRI scans and the tracking system used to calculate the location and position of the tumor are both FDA approved technologies.

The research doctors will also use the MRI scans to evaluate any changes in your lung function during and following your radiation treatments.

In this study the participant will undergo a series of MRI scans with and without contrast dye.

This study is being funded through grants from the National Institutes of Health (NIH).

DETAILED DESCRIPTION:
In this protocol, we seek to assess whether tumor motion can be inferred using dynamic MRI and external surrogates. We propose to (1) investigate the feasibility of tracking the real-time tumor position using dynamic MRI and inferring tumor position using external surrogates placed on the skin of the subject and (2) determine lung function during and following radiation by assessing lung perfusion maps obtained via dynamic MRI with dose maps in order to determine image-based biomarkers for lung toxicity following radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years old or older
* Patients must be undergoing radiation therapy with or without chemotherapy for thoracic and/or abdominal cancers.

Exclusion Criteria:

* Pregnant or breast-feeding women are excluded. Negative serum or urine pregnancy test prior to study entry is required. Once on the protocol, the patient will be advised and expected to implement an accepted and effective method of contraception such as oral contraceptives (birthcontrol pill), intrauterine devices (IUDs), contraceptive implants under skin or contraceptive injections and condoms with foam.
* Patients with kidney disease of any severity or on hemodialysis.
* Patients who have metallic dental fillings or other metallic implants.
* Patients with known allergies to gadolinium-based contrast agents.
* Patients who have difficulty lying flat on their back for extended periods of time will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients must be undergoing radiation therapy with or without chemotherapy for thoracic and/or abdominal cancers.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2009-11; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Warren D. D'Souza, PhD, Principal Investigator — UMMC MSGCC Department of Radiation Oncology
Locations (1):
- Ummc Msgcc, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Dynamic Lung MRI: Lung Tumor Motion and Function
Period: Overall Study
Arm/Group | Dynamic Lung MRI
Started | 16
Completed | 7
Not Completed | 9

BASELINE CHARACTERISTICS:
Groups:
- Dynmaic Lung MRI: Lung Tumor Motion and Function
Arm/Group | Dynmaic Lung MRI
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Whose Tumor Position is Visible Within ~2mm Using Cine-MRI Scans and External Sensors
Description: Tumor tracking using cine-MRI and external surrogates with an accuracy of ~ 2mm.
  The participants' tumor size/margins were not specficially defined as long as it was visible/measurable on the MRI.
Time Frame: 2 years
Measure: Number; unit: participants
Groups:
- Lung Tumor Motion and Lung Function: This is a pilot study and there is only one group.
Arm/Group | Lung Tumor Motion and Lung Function
Number analyzed (Participants) | 16
participants | 7

2. Secondary Outcome: Number of Participants Whose Tumor Motion Could be Tracked Using Dynamic MRI w/ Contrast Post Radiation
Description: The internal margin (IM) is one half of the peak-to-peak displacement amplitude on 4D-CT images.
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Dynamic Lung MRI
Number analyzed (Participants) | 16
participants | 7

ADVERSE EVENTS:
Arm/Group | Dynamic Lung MRI
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes